CLINICAL TRIAL: NCT03462628
Title: Additional Low Voltage Area Ablation in Older Patients With Paroxysmal Atrial Fibrillation: a Randomized Control Trial of STABLE-SR-III
Brief Title: Additional Low Voltage Area Ablation in Older Patients With Paroxysmal Atrial Fibrillation
Acronym: STABLE-SR-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other); First Affiliated Hospital of Wannan Medical College (Other); Second Affiliated Hospital of Nantong University (Other); Zhongda Hospital (Other); The Third Affiliated Hospital of Soochow University (Other); The Second Hospital of Hebei Medical University (Other); The First Affiliated Hospital of Soochow University (Other); Xuzhou Central Hospital, the Affiliated Xuzhou Hospital of Medical College of Southeast University (Unknown); Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Minglong Chen, Deputy Director of the Department of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-SR-085
Record Dates: First submitted 2018-03-01; First posted 2018-03-12 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: substrate modification; pulmonary vein isolation; ablation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): PVI with additional low-voltage substrate modification
  Interventions: Procedure: CPVI plus low-voltage substrate modification
- Control Group (Active Comparator): PVI only
  Interventions: Procedure: CPVI alone

INTERVENTIONS:
Procedure: CPVI plus low-voltage substrate modification — CPVI plus low-voltage substrate modification in the left atrium during SR
  Other Names: CPVI plus additional low-voltage substrate modification
  Arms: Study Group
Procedure: CPVI alone — circumferential pulmonary vein isolation
  Arms: Control Group

SUMMARY:
The primary objective of this investigation is to compare the efficacy of two different AF ablation strategies in older patients with paroxysmal AF: Pulmonary vein isolation alone versus additional low-voltage substrate modification during sinus rhythm

DETAILED DESCRIPTION:
BACKGROUND: Atrial fibrillation (AF) is the most common cardiac rhythm disorder. Catheter ablation to the pulmonary veins isolation (PVI) electrically from the left atrium (LA) has been shown to be an effective treatment for paroxysmal AF (PAF). The consensus is that PVI alone is the main strategy for PAF ablation. Based on the results from our pilot study and STABLE-SR trial, that low-voltage modification beyond CPVI is very promising for persistent AF ablation. Whether the low voltage area modification combined with PVI improves outcomes is unclear in older patients with PAF.

AIM OF THE STUDY: The primary objective of this investigation is to compare the efficacy of two different AF ablation strategies in older patients with PAF: PVI alone versus additional low-voltage substrate modification during sinus rhythm. The primary endpoint is freedom from AF and/or ATs with or without antiarrhythmic drugs (AADs) at 12 months after a single-ablation procedure. AF and/or AT occurring in the first 3 months after the ablation (blanking period) was censored. Each atrial tachyarrhythmia episode lasts > 30 seconds monitored by ECG, 24-Holter or 7 days-Holter was defined as recurrence. The secondary endpoint are incidence of periprocedural complications, including stroke, PV stenosis, cardiac perforation, esophageal injury and death; procedure time; fluoroscopy time (including the total fluoroscopy time, during CPVI and after CPVI); the occurrence of the conversion from AF to AT, and its relationship with long-term outcome; the scar distribution and the relationship of success rate in older PAF patients.

STUDY DESIGN: This is a randomized, prospective, parallel, single-blind multicenter design. The expected freedom from atrial fibrillation in older patients after one ablation procedure was 75% for PVI. Previous study did not include a group assigned to isolation plus additional low-voltage substrate modification during sinus rhythm, so freedom form AF for this procedure was estimated from the literature at 85%. A log-rank test was used for sample-size calculation. To test whether the isolation plus low-voltage substrate modification was superior to isolation only. Then the 369 patients were needed, with a randomization ratio of 1:1, for the study to have a power of 90% at a two-sided alpha level of 0.05. Assuming a dropout rate of 15%, we need 434 patients. Patients are randomized in a 1:1 fashion into one of the investigation arms: CPVI plus low-voltage substrate modification in the left atrium during SR and CPVI alone. Follow-up for these patients includes visits at 3 m, 6 m, 9 m, 12 m.

ELIGIBILITY:
Inclusion Criteria:

* Patients age is 65-80 years;
* Patients with paroxysmal AF;
* Patients can sign the written informed consent for the study;
* Patients can endure the required follow-up.

Exclusion Criteria:

* Patients with previous radiofrequency ablation;
* Patients with PLT count less than 80×109/L, or with contraindications to systemic anticoagulation with heparin or Coumadin or a direct thrombin inhibitor;
* Patients with left atrial size ≥ 55 mm (2D echocardiography, parasternal long-axis view);
* Patients with thromboemboli in LA (TEE or MSCT);
* Patients with severe structural cardiac disease (medium or severe mitral regurgitation, DCM, HCM, or other severe valvular heart diseases);
* Patients with abnormal thyroid function;
* Patients with severe liver or renal dysfunction (AST or ALT > 3-fold of upper limit value; the SCr > 3.5 mg/dl or Ccr < 30 ml/min);
* Previous surgery history in last 3 months;
* Patients with life expectancy < 12 months

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 438 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Freedom from AF and/or ATs with or without antiarrhythmic drugs (AADs) | at least 12 months follow up]
  Freedom from AF and/or ATs with or without antiarrhythmic drugs (AADs) at 12months after a single-ablation procedure. AF and/or AT occurring in the first 3 months after the ablation (blanking period) was censored. Each episode lasts > 30 seconds.

SECONDARY OUTCOMES:
Incidence of peri-procedural complications | 1 week after patient enrollment
  stroke, cardiac perforation, and death
complications during the follow-up | 1month to 12 months
  PV stenosis, esophageal injury
Procedure time | 1 week after patient enrollment
  time that the patient spend in the procedure room
Fluoroscopy time | 1 week after patient enrollment
  the total fluoroscopy time, during PVI alone or PVI plus low-voltage substrate modification

CONTACTS AND LOCATIONS:
Overall Officials: Minglong Chen, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, China

REFERENCES:
- [Derived] Qi X, Chen H, Yang G, Liu H, Wang Z, Jiang X, Cui C, Cai C, Ju W, Chen M. Unipolar Voltage for Better Characterizing Left Atrium Substrates: Comparing the Predictive Efficacy for Recurrence Post Atrial Fibrillation Ablation in a Post Hoc Analysis of STABLE-SR-III Trial. J Cardiovasc Electrophysiol. 2025 Jan;36(1):149-156. doi: 10.1111/jce.16490. Epub 2024 Nov 7. PMID 39511789
- [Derived] Chen H, Li C, Han B, Xiao F, Yi F, Wei Y, Jiang C, Zou C, Shi L, Ma W, Wang W, Wang Y, Du H, Chen L, Chen M; STABLE-SR-III Investigators. Circumferential Pulmonary Vein Isolation With vs Without Additional Low-Voltage-Area Ablation in Older Patients With Paroxysmal Atrial Fibrillation: A Randomized Clinical Trial. JAMA Cardiol. 2023 Aug 1;8(8):765-772. doi: 10.1001/jamacardio.2023.1749. PMID 37378966